CLINICAL TRIAL: NCT05009277
Title: Study To Evaluate The Sensitivity Of The Linda Thermal Device In Relation To Mammography In The Detection Of Suspected Breast Neoplasia
Brief Title: Study To Evaluate The Sensitivity Of The Linda Thermal Device
Acronym: LINDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Termo Health Tecnologia Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: LINDA
Record Dates: First submitted 2021-06-08; First posted 2021-08-17 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Device; Thermography; Mammography
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Device — LINDA thermal device
  Other Names: LINDA

SUMMARY:
The LINDA thermal device consists of a thermal camera attachable to a cell phone and an application for connection with an artificial intelligence program based on a convolutional neural network for classification of thermographic breast images. The system is previously fed with thermographic images of the breast and their respective results/diagnostics. The images are processed in an automated way and return a percentage of chance of having a pathological pattern.

DETAILED DESCRIPTION:
The LINDA thermal device consists of a thermal camera attachable to a cell phone and an application for connection with an artificial intelligence program based on a convolutional neural network for classification of thermographic breast images. The system is previously fed with thermographic images of the breast and their respective results/diagnostics. The images are processed in an automated way and return a percentage of chance of having a pathological pattern.

nfrared imaging (thermography) was approved as an auxiliary imaging modality for mammography by the Food and Drug Administration (FDA) in 1982. Thermography is a non-invasive, non-contact method without ionizing radiation, which is why its use can be prolonged and repeated. This technique allows for an evaluation of the functionality of the structures, which is why it is considered a physiological test and records the variation in the surface temperature of the human body based on the infrared radiation emitted by the surface of that body. It is capable of detecting tumor lesions since cancer cells generate heat due to the release of nitric oxide in the blood, causing changes in microcirculation, vasodilation, neo-angiogenesis and increased metabolic activity of cancer cells. Thus, in the initial stage of breast cancer, when it has not yet caused anatomical changes, there will be physiological changes that will lead to an increase in blood flow and metabolic activity. This increase induces a temperature rise in the area which will then be detected by thermography.

ELIGIBILITY:
Inclusion Criteria:

1. Provide your signed and dated consent in duplicate;
2. Female, aged between 40 and 69 years;
3. Have had a mammography no more than 6 months before V1 and with results available in V1.

Exclusion Criteria:

1. Fever (temperature above 37.8°C at rest) in the last 48 hours before image capture by thermography;
2. Exposure to natural or artificial light for chest tanning for less than three (3) days before performing the thermography;
3. Pregnant or breastfeeding women in the last 6 months;
4. Physical exercise 3 h before performing the thermography;
5. To have performed a breast biopsy less than 6 months after the thermography;
6. Other conditions that, at the investigator's discretion, increase the risk to the patient or make her unsuitable for the study.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study population will be composed of female subjects between 40 and 69 years of age, which has performed a mammography during the past 6 months before inclusion and that has the result available and is willing to consent to have image captured via thermographic camera.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
assess thermal sensitivity | assess thermal sensitivity immediatly after capturing the image
  The primary objective of the study is to assess the thermal sensitivity of the LINDA device in detecting suspected breast cancer compared to mammography.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens F Mendrone, Study Chair — Termo Health Tecnologia Ltda
Locations (1):
- Hospital Vera Cruz, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.